CLINICAL TRIAL: NCT00856219
Title: Comparison of Enteral Versus Parenteral Feeding in Healthy Human Subjects
Acronym: Feeding
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0220044983
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Immune System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enteral Continuous (Active Comparator): Continuous tube feeding for 72 hours.
  Interventions: Dietary Supplement: Enteral Continuous
- Enteral Intermittent (Active Comparator): Intermittent tube feedings for 72 hours
  Interventions: Dietary Supplement: Enteral Intermittent
- Parenteral (Active Comparator): Parenteral continuously for 72 hours
  Interventions: Dietary Supplement: Parenteral Continuous

INTERVENTIONS:
Dietary Supplement: Enteral Continuous — Continuous Tube Feeding for 72 hours
  Arms: Enteral Continuous
Dietary Supplement: Enteral Intermittent — Intermittent Tube Feedings
  Arms: Enteral Intermittent
Dietary Supplement: Parenteral Continuous — Parenteral Continuously for 72 hours
  Arms: Parenteral

SUMMARY:
Literature suggests that route of feeding and/or certain nutrients may cause alterations in the body's immune cells. Immune cells help protect the body and fight infection/disease. Tube feeding (TF) is a method of delivering nutrition directly to the stomach/intestines via a small tube. The immune system may respond differently when receiving continuous TF as compared to receiving intermittent TF. Heart rate variability (HRV, the intervals between heartbeats) is a measurement of the nervous system's response to a stress/illness. The differences in immune cells and/or HRV may influence how the body reacts to complications such as infection.

ELIGIBILITY:
Inclusion Criteria:

* General good health as demonstrated by medical history, physical& laboratory tests
* Age between 18 and 40 years
* Written informed consent prior to the performance of any study related procedures

Exclusion Criteria:

* History of cancer, rheumatoid arthritis, or immunological, renal, hepatic, endocrine, neurologic, heart disease or hypertension
* Any medication taken in past 48 hrs (except birth control)
* Recent history of alcohol or drug abuse
* Unable to provide written informed consent
* Exposure to any experimental agent or procedure within 30 days of study
* Pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Route and type of feeding on Immune response | Day 1- Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Corbett, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Rutgers-RWJMS, New Brunswick, New Jersey, United States